CLINICAL TRIAL: NCT00404820
Title: A Multi-center, Randomized, Open-label, Controlled, One-year Trial to Measure the Effect of Zoledronic Acid and Alendronate on Bone Metabolism in Postmenopausal Women With Osteopenia and Osteoporosis
Brief Title: Safety/Efficacy of Zoledronic Acid and Alendronate on Bone Metabolism in Postmenopausal Women With Osteoporosis
Acronym: ROSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446HDE31
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Osteoporosis
Keywords: osteoporosis; bisphosphonate; biomarker; zoledronic acid; alendronate; postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid; Solutions; Alendronate; Calcium; Vitamin D

ARMS (2):
- Zoledronic acid 5 mg (Experimental): Patients received zoledronic acid 5 mg in 100 ml solution in a 15 minute intravenous (iv) infusion once per year. The peripheral iv infusion was preceded by and followed by a 10 ml normal saline flush of the intravenous line. In addition to study therapy, all participants received 1200 mg elemental calcium and 800 IU of vitamin D daily. Calcium and vitamin D were supplied in a chewable tablet that was to be taken twice daily.
  Interventions: Drug: Zoledronic acid 5 mg solution; Drug: Calcium/Vitamin D
- Alendronate 70 mg (Active Comparator): Patients received an alendronate 70 mg tablet once weekly with 200 ml of tap water in the morning on an empty stomach at least 30 minutes before the first meal. Patients were to remain in an upright position for 30 minutes after swallowing the tablet. In addition to study therapy, all participants received 1200 mg elemental calcium and 800 IU of vitamin D daily. Calcium and vitamin D were supplied in a chewable tablet that was to be taken twice daily.
  Interventions: Drug: Alendronate 70 mg tablets; Drug: Calcium/Vitamin D

INTERVENTIONS:
Drug: Zoledronic acid 5 mg solution — Zoledronic acid was supplied as a concentrate of 5.33 mg zoledronic acid monohydrate in a 100 ml solution. 5.33 mg zoledronic acid monohydrate equals 5 mg zoledronic acid.
  Arms: Zoledronic acid 5 mg
Drug: Alendronate 70 mg tablets — Patients received an alendronate 70 mg tablet once weekly with 200 ml of tap water in the morning on an empty stomach at least 30 minutes before the first meal.
  Arms: Alendronate 70 mg
Drug: Calcium/Vitamin D — Combined elemental calcium / vitamin D chewable tablets. Participants took 2 tablets a day, for a daily dose of calcium 1200 mg/vitamin D 800 IU.

SUMMARY:
The aim of this study was to examine the effect of zoledronic acid and alendronate on bone metabolism as measured by biomarkers in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

- Low bone mineral density (as indicated by a "t-score" of -2.0 or lower) postmenopausal women

Exclusion Criteria:

- Previous use of oral and iv bisphosphonates, parathormone, strontium ranelate, sodium fluoride.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma GmbH, Germany +49 911 273-0, Study Director — Novartis
Locations (1):
- For site information contact Novartis Pharmaceuticals, Multiple Cities, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Germany; first patient enrolled October 2006 and completed December 2008.
Period: Overall Study
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Started | 408 | 196
Started Treatment | 408 | 194 (The reason why 2 patients did not start treatment is unavailable.)
Completed | 389 | 172
Not Completed | 19 | 24
Not completed — Adverse Event | 4 | 16
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 7 | 3
Not completed — Administrative problems | 2 | 0
Not completed — Death | 1 | 0
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg | Total
Number analyzed (Participants) | 408 | 194 | 602
Age Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.1) | 68.2 (7.9) | 67.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 408 | 194 | 602
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Cross-linked N-telopeptide of Type I Collagen (NTx) Level Assessed as Standardized Area Under the Curve From Screening to Month 12 in the Intent-to-Treat Population
Description: The level of bone activity as measured by NTx over the course of 12 months was assessed using the standardized area under the curve. Blood samples were collected after an overnight fast of at least 8 hours between 7:00 and 11:00 AM at Screening and Months 1.5, 3, 6, 9, and 12 months after baseline. Serum was analyzed at a central lab using commercially available ELISA kits. Standardized AUC was calculated by the AUC divided by the number of days the patient participated in the study.
Time Frame: Screening to end of study (Month 12)
Population: Intent-to-treat sample (ITT) population: All patients who received at least 1 dose of study medication and who had at least 1 post-baseline determination of cross-linked N-telopeptide of type I collagen (NTx) level.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Number analyzed (Participants) | 408 | 191
ng/ml | 0.282 (0.195) | 0.270 (0.266)

2. Secondary Outcome: Change of Procollagen Type I Nitrogenous Propeptide (P1NP) Level Assessed as Standardized Area Under the Curve From Screening to Month 12
Description: The level of bone activity as measured by P1NP over the course of 12 months was assessed using the standardized area under the curve. Blood samples were collected after an overnight fast of at least 8 hours between 7:00 and 11:00 AM at Screening and Months 1.5, 3, 6, 9, and 12 months after baseline. Serum was analyzed at a central lab using commercially available ELISA kits. Standardized AUC was calculated by the AUC divided by the number of days the patient participated in the study.
Time Frame: Screening to end of study (Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Number analyzed (Participants) | 408 | 191
ng/ml | 28.2 (23.0) | 25.5 (17.6)

3. Secondary Outcome: Change in the Qualeffo-41 Quality of Life (QoL) Questionnaire Score From Baseline to Month 12
Description: The Qualeffo-41 QoL questionnaire was completed by the patient at Baseline and at Month 12. The questionnaire includes 41 questions covering 7 domains (pain, physical function and activities of daily living, physical function and jobs around the house, physical function and mobility, leisure and social activities, general health perception, mental function). Scores on each question range from 1 to 3, 4, or 5. The total score summed over all questions ranges from 41-205 points; the lower the score the higher the quality of life. A negative change score indicates improvement.
Time Frame: Baseline to end of study (Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Number analyzed (Participants) | 408 | 191
Units on a scale | -1.2 (8.8) | -0.6 (9.0)

4. Secondary Outcome: Number of Patients With a Clinical Fracture From Baseline to Month 12
Description: A diagnosis of clinical fracture was based on physical examination findings, ie, swelling, tenderness, limited movement, pain.
Time Frame: Baseline to end of study (Month 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Number analyzed (Participants) | 408 | 191
Participants | 10 | 4

5. Secondary Outcome: Change in Body Height From Baseline to Month 12
Description: Body height was measured at Baseline and at the end of the study (Month 12) and the change in height calculated.
Time Frame: Baseline to end of study (Month 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Number analyzed (Participants) | 408 | 191
cm | -0.1 (1.0) | 0.0 (1.2)

6. Secondary Outcome: Therapy Preference at End of Study (Month 12)
Description: Patients were administered a questionnaire at the end of the study in which they were asked which type of therapy, weekly oral or yearly iv, they preferred.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Number analyzed (Participants) | 408 | 191
Participants
  No data available | 30 | 16
  Yearly iv | 330 | 82
  Weekly oral | 48 | 93

7. Primary Outcome: Change of Cross-linked N-telopeptide of Type I Collagen (NTx) Level Assessed as Standardized Area Under the Curve From Screening to Month 12 in the Per Protocol Population
Description: as for outcome 1
Time Frame: Screening to end of study (Month 12)
Population: Per Protocol population: All intent-to-treat patients who did not show major deviations from the protocol procedures that may have had an impact on the study outcome.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Number analyzed (Participants) | 349 | 146
ng/ml | 0.293 (0.199) | 0.294 (0.175)

ADVERSE EVENTS:
Arm/Group | Zoledronic Acid 5 mg | Alendronate 70 mg
Serious Adverse Events (participants affected / at risk) | 43/408 | 21/194
Other Adverse Events (participants affected / at risk) | 267/408 | 94/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 5 mg (N=408) | Alendronate 70 mg (N=194)
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Visual disturbance (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
C-Reactive protein increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular vascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lo of consciousness (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Presenile dementia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Uterine cyst (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial bypass operation (Surgical and medical procedures) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 3
Femoral artery occlusion (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 5 mg (N=408) | Alendronate 70 mg (N=194)
Abdominal pain upper (Gastrointestinal disorders) | 12 | 13
Constipation (Gastrointestinal disorders) | 9 | 10
Diarrhoea (Gastrointestinal disorders) | 9 | 10
Dyspepsia (Gastrointestinal disorders) | 3 | 14
Nausea (Gastrointestinal disorders) | 23 | 11
Fatigue (General disorders) | 24 | 4
Influenza like illness (General disorders) | 132 | 5
Pyrexia (General disorders) | 21 | 2
Nasopharyngitis (Infections and infestations) | 26 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 52 | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 23 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 5
Headache (Nervous system disorders) | 43 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.